CLINICAL TRIAL: NCT04342507
Title: Effects of Probiotic Oral Supplementation on the Treatment of Chalazion in Adults: a Pilot Study on 20 Patients
Brief Title: Probiotics for Treatment of Chalazion in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08/2019
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Chalazion
Keywords: microbiome/microbiota; probiotics; adults
MeSH Terms: conditions — Chalazion | interventions — Conservative Treatment; Probiotics

STUDY DESIGN:
Intervention Model Description: Prospective comparative pilot study with two groups randomly divided
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: conservative (Other): conservative treatment with lid hygiene, warm compression, and dexamethasone/tobramycin ointment for at least 20 days
  Interventions: Other: conservative treatment
- Group B: probiotics (Experimental): in addition to the conservative treatment they receive probiotics mixture (Streptococcus thermophilus, Lactococcus lactis, Lactobacillus delbrueckii subsp. bulgaricus) once a day up to 3 months.
  Interventions: Other: conservative treatment; Dietary Supplement: probiotics

INTERVENTIONS:
Other: conservative treatment — lid hygiene, warm compression, and dexamethasone/tobramycin ointment for at least 20 days.
Dietary Supplement: probiotics — use specific probiotics in addiction to conservative treatment to modify the intestinal microbiome to ameliorate the clinical course of adults chalazia by re-establishing intestinal and immune homeostasis
  Arms: Group B: probiotics

SUMMARY:
There is growing evidence encouraging probiotics use in several diseases. The aim of the investigator's study is to define the possible beneficial impact of probiotics on adults suffering from chalazia.

DETAILED DESCRIPTION:
Prospective comparative pilot study on 20 adults suffering from chalazion randomly divided into two groups. The first group, received conservative treatment with lid hygiene, warm compression, and dexamethasone/tobramycin ointment for at least 20 days. The second group, in addition to the conservative treatment, received a mixture of probiotic microorganisms once a day up to 3 months. Chalazia were classified according to their size into three groups: small (≤2 mm), medium (2-4 mm), or large (>4 mm). When conservative treatment (with and without probiotics supplementation) failed to resolve the lesion, invasive methods were used, (intralesion steroid injection in medium size chalazion and surgical incision and curettage for the largest ones).

ELIGIBILITY:
Inclusion Criteria:

* history of rapid onset of painful inflamed mass that had reached a stationary size for more than 2 months
* clinical appearance and location of the lesion

Exclusion Criteria:

* eyelid infection
* chalazion duration < 1 month
* nonpalpable chalazion
* suspicion of malignancy
* comorbidities (constitutional atopy and seborrheic dermatitis, hormonal dysfunction, presence of irritable bowel disease, infectious mainly related to Staphylococcus aureus and Propionibacterium acnes, demodex mite infestation, vitamin A deficiency, arterial hypertension, diabetes and pregnancy)
* personal habits (smoking, eating disorders, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
healing time | 3 months
  healing time changes with a complete resolution of chalazion

SECONDARY OUTCOMES:
recurrences | six months
  evaluation of recurrences in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, Full Professor, Principal Investigator — University of Molise
Locations (1):
- University of Molise, Campobasso, Molise, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gilchrist H, Lee G. Management of chalazia in general practice. Aust Fam Physician. 2009 May;38(5):311-4. PMID 19458801
- [Result] Unal M. Chalazion treatment. Orbit. 2008;27(6):397-8. doi: 10.1080/01676830802623174. No abstract available. PMID 19085290
- [Result] Sklar BA, Gervasio KA, Leng S, Ghosh A, Chari A, Wu AY. Management and outcomes of proteasome inhibitor associated chalazia and blepharitis: a case series. BMC Ophthalmol. 2019 May 14;19(1):110. doi: 10.1186/s12886-019-1118-x. PMID 31088416
- [Result] Nemet AY, Vinker S, Kaiserman I. Associated morbidity of chalazia. Cornea. 2011 Dec;30(12):1376-81. doi: 10.1097/ICO.0b013e31821de36f. PMID 21993469
- [Result] Yam JC, Tang BS, Chan TM, Cheng AC. Ocular demodicidosis as a risk factor of adult recurrent chalazion. Eur J Ophthalmol. 2014 Mar-Apr;24(2):159-63. doi: 10.5301/ejo.5000341. Epub 2013 Jul 16. PMID 23873491
- [Result] Burkhart CG, Burkhart CN. Similar to acne vulgaris, bacteria may produce the biological glue that causes plugging of the meibomian gland leading to chalazions. Clin Exp Ophthalmol. 2008 Apr;36(3):295; author reply 295-6. doi: 10.1111/j.1442-9071.2008.01714.x. No abstract available. PMID 18412605
- [Result] Malekahmadi M, Farrahi F, Tajdini A. Serum Vitamin A Levels in Patients with Chalazion. Med Hypothesis Discov Innov Ophthalmol. 2017 Fall;6(3):63-66. PMID 29392144
- [Result] Nabie R, Soleimani H, Nikniaz L, Raoufi S, Hassanpour E, Mamaghani S, Bahremani E. A prospective randomized study comparing incision and curettage with injection of triamcinolone acetonide for chronic chalazia. J Curr Ophthalmol. 2019 May 7;31(3):323-326. doi: 10.1016/j.joco.2019.04.001. eCollection 2019 Sep. PMID 31528769
- [Result] Lee JW, Yau GS, Wong MY, Yuen CY. A comparison of intralesional triamcinolone acetonide injection for primary chalazion in children and adults. ScientificWorldJournal. 2014;2014:413729. doi: 10.1155/2014/413729. Epub 2014 Oct 15. PMID 25386597
- [Result] Kerry RG, Patra JK, Gouda S, Park Y, Shin HS, Das G. Benefaction of probiotics for human health: A review. J Food Drug Anal. 2018 Jul;26(3):927-939. doi: 10.1016/j.jfda.2018.01.002. Epub 2018 Feb 2. PMID 29976412
- [Result] Han KJ, Lee JE, Lee NK, Paik HD. Antioxidant and Anti-Inflammatory Effect of Probiotic Lactobacillus plantarum KU15149 Derived from Korean Homemade Diced-Radish Kimchi. J Microbiol Biotechnol. 2020 Apr 28;30(4):591-598. doi: 10.4014/jmb.2002.02052. PMID 32238771
- [Result] Morrison DJ, Preston T. Formation of short chain fatty acids by the gut microbiota and their impact on human metabolism. Gut Microbes. 2016 May 3;7(3):189-200. doi: 10.1080/19490976.2015.1134082. Epub 2016 Mar 10. PMID 26963409
- [Result] Kalyana Chakravarthy S, Jayasudha R, Sai Prashanthi G, Ali MH, Sharma S, Tyagi M, Shivaji S. Dysbiosis in the Gut Bacterial Microbiome of Patients with Uveitis, an Inflammatory Disease of the Eye. Indian J Microbiol. 2018 Dec;58(4):457-469. doi: 10.1007/s12088-018-0746-9. Epub 2018 Jun 4. PMID 30262956
- [Result] Iovieno A, Lambiase A, Sacchetti M, Stampachiacchiere B, Micera A, Bonini S. Preliminary evidence of the efficacy of probiotic eye-drop treatment in patients with vernal keratoconjunctivitis. Graefes Arch Clin Exp Ophthalmol. 2008 Mar;246(3):435-41. doi: 10.1007/s00417-007-0682-6. Epub 2007 Nov 27. PMID 18040708
- [Result] Tavakoli A, Flanagan JL. The Case for a More Holistic Approach to Dry Eye Disease: Is It Time to Move beyond Antibiotics? Antibiotics (Basel). 2019 Jun 30;8(3):88. doi: 10.3390/antibiotics8030088. PMID 31262073
- [Result] Lin P. The role of the intestinal microbiome in ocular inflammatory disease. Curr Opin Ophthalmol. 2018 May;29(3):261-266. doi: 10.1097/ICU.0000000000000465. PMID 29538183
- [Result] Baim AD, Movahedan A, Farooq AV, Skondra D. The microbiome and ophthalmic disease. Exp Biol Med (Maywood). 2019 Apr;244(6):419-429. doi: 10.1177/1535370218813616. Epub 2018 Nov 21. PMID 30463439
- [Result] Cavuoto KM, Banerjee S, Galor A. Relationship between the microbiome and ocular health. Ocul Surf. 2019 Jul;17(3):384-392. doi: 10.1016/j.jtos.2019.05.006. Epub 2019 May 21. PMID 31125783
- [Result] Lin P. Importance of the intestinal microbiota in ocular inflammatory diseases: A review. Clin Exp Ophthalmol. 2019 Apr;47(3):418-422. doi: 10.1111/ceo.13493. Epub 2019 Mar 25. PMID 30834680
- [Result] Nelson JD, Shimazaki J, Benitez-del-Castillo JM, Craig JP, McCulley JP, Den S, Foulks GN. The international workshop on meibomian gland dysfunction: report of the definition and classification subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1930-7. doi: 10.1167/iovs.10-6997b. Print 2011 Mar. No abstract available. PMID 21450914
- [Result] Ozdal PC, Codere F, Callejo S, Caissie AL, Burnier MN. Accuracy of the clinical diagnosis of chalazion. Eye (Lond). 2004 Feb;18(2):135-8. doi: 10.1038/sj.eye.6700603. PMID 14762403
- [Result] Ozkan J, Willcox MD. The Ocular Microbiome: Molecular Characterisation of a Unique and Low Microbial Environment. Curr Eye Res. 2019 Jul;44(7):685-694. doi: 10.1080/02713683.2019.1570526. Epub 2019 Feb 4. PMID 30640553
- [Result] Wen X, Miao L, Deng Y, Bible PW, Hu X, Zou Y, Liu Y, Guo S, Liang J, Chen T, Peng GH, Chen W, Liang L, Wei L. The Influence of Age and Sex on Ocular Surface Microbiota in Healthy Adults. Invest Ophthalmol Vis Sci. 2017 Dec 1;58(14):6030-6037. doi: 10.1167/iovs.17-22957. PMID 29196767
- [Result] Grzybowski A, Brona P, Kim SJ. Microbial flora and resistance in ophthalmology: a review. Graefes Arch Clin Exp Ophthalmol. 2017 May;255(5):851-862. doi: 10.1007/s00417-017-3608-y. Epub 2017 Feb 22. PMID 28229218
- [Result] Lu LJ, Liu J. Human Microbiota and Ophthalmic Disease. Yale J Biol Med. 2016 Sep 30;89(3):325-330. eCollection 2016 Sep. PMID 27698616
- [Result] Rosenbaum JT, Lin P, Asquith M. The microbiome, HLA, and the pathogenesis of uveitis. Jpn J Ophthalmol. 2016 Jan;60(1):1-6. doi: 10.1007/s10384-015-0416-y. Epub 2015 Sep 14. PMID 26370944
- [Result] Nayyar A, Gindina S, Barron A, Hu Y, Danias J. Do epigenetic changes caused by commensal microbiota contribute to development of ocular disease? A review of evidence. Hum Genomics. 2020 Mar 13;14(1):11. doi: 10.1186/s40246-020-00257-5. PMID 32169120
- [Result] Verhagen FH, Bekker CPJ, Rossato M, Hiddingh S, de Vries L, Devaprasad A, Pandit A, Ossewaarde-van Norel J, Ten Dam N, Moret-Pot MCA, Imhof SM, de Boer JH, Radstake TRDJ, Kuiper JJW. A Disease-Associated MicroRNA Cluster Links Inflammatory Pathways and an Altered Composition of Leukocyte Subsets to Noninfectious Uveitis. Invest Ophthalmol Vis Sci. 2018 Feb 1;59(2):878-888. doi: 10.1167/iovs.17-23643. PMID 29435587
- [Result] Forbes JD, Chen CY, Knox NC, Marrie RA, El-Gabalawy H, de Kievit T, Alfa M, Bernstein CN, Van Domselaar G. A comparative study of the gut microbiota in immune-mediated inflammatory diseases-does a common dysbiosis exist? Microbiome. 2018 Dec 13;6(1):221. doi: 10.1186/s40168-018-0603-4. PMID 30545401
- [Result] Trujillo-Vargas CM, Schaefer L, Alam J, Pflugfelder SC, Britton RA, de Paiva CS. The gut-eye-lacrimal gland-microbiome axis in Sjogren Syndrome. Ocul Surf. 2020 Apr;18(2):335-344. doi: 10.1016/j.jtos.2019.10.006. Epub 2019 Oct 20. PMID 31644955
- [Result] Kugadas A, Wright Q, Geddes-McAlister J, Gadjeva M. Role of Microbiota in Strengthening Ocular Mucosal Barrier Function Through Secretory IgA. Invest Ophthalmol Vis Sci. 2017 Sep 1;58(11):4593-4600. doi: 10.1167/iovs.17-22119. PMID 28892827
- See also: MicroRNAs and microbiota: Is there a cross talk? — https://journals.prous.com/journals/servlet/xmlxsl/pk_journals.xml_summary_pr?p_JournalId=4&p_RefId=3079409&p_IsPs=N